CLINICAL TRIAL: NCT03483701
Title: Cognitive Remediation Therapy for Patients With Serious Mental Illness Who Failed to Benefit From Supported Employment
Brief Title: Thinking Skills at Work: Cognitive Remediation Therapy for Patients With Serious Mental Illness
Acronym: TSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: Ministry of Social Development and Poverty Reduction, British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHREB No. 2016-096
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia and Related Disorders; Psychotic Disorder
Keywords: Cognitive Remediation Therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This randomized controlled trial will use a single-blind study design with two treatment arms. The research team that assesses participants at baseline and follow-up will have no knowledge of their assigned treatment arm. The participants, however, will know which treatment arm they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation Therapy (Experimental): Participants in the experimental group will continue to receive IPS services, which is part of their standard care. In addition, they will be required to complete up to 5 hours per week of computerized cognitive exercises. Cognitive training can be done at home on a computer, on their own schedule. Participants will also receive 1 hour/week of individual coaching to discuss cognitive remediation progress, learn about different cognitive domains and develop ways to generalize their cognitive remediation gains.
  Interventions: Behavioral: Cognitive Remediation Therapy
- Treatment as Usual (No Intervention): Participants in the control condition will continue to receive IPS services as usual.

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — The intervention of interest for participants in the experimental group is the addition of up to 5 hours per week of computerized cognitive exercises. Cognitive training can be done at home on a computer. For participants without access to a computer, a laptop/tablet computer with the necessary software will be provided for the duration of training. Participants will be able to complete the cognitive exercises on their own schedule, with participation verified by the software. Participants will also receive 1 hour/week of individual coaching to discuss cognitive remediation progress, e.g. to learn about different cognitive domains and develop ways to generalize their cognitive remediation gains.
  Arms: Cognitive Remediation Therapy

SUMMARY:
The purpose of this study is to help people with serious mental illness get and keep the job they want by improving their thinking skills, using cognitive remediation therapy. For people with serious mental illness, the Individual Placement and Support (IPS) Program is an effective approach to help people become employed. Despite its general success, still only 55% of clients find employment. Most of that success occurs in the first three months; after six months, the chances of finding competitive work are quite low. Among those who fail to find employment with IPS, cognitive dysfunction is often a significant problem. The proposed study will target IPS clients who have not found work after 3 months of employment-support services: our hypothesis is that, after three months with no success, the addition of cognitive remediation to IPS will improve employment rates (compared to those who continue to receive IPS alone).

The proposed randomized controlled trial will use a single-blind study design, focused on IPS clients who are slow to (or may never) find employment success. Specifically, the proposed study will have two treatment arms: a) cognitive remediation added to continued IPS services, and b) continued IPS services alone. The study will collaborate with IPS workers at 11 Mental Health and Substance Use (MHSU) clinics to identify clients who are non-responders in the first 3 months, and seek their consent to participate in the study. They will be randomized to either TAU (continuation with IPS and other standard treatments), or TAU plus cognitive remediation. The CRT will consist of computerized cognitive exercise practice, strategy coaching, and teaching coping/compensatory strategies for 12 weeks. Clients will be assessed at 3-time points: prior to the start of cognitive remediation ("baseline"), end-point (3-month), and 6 months after the endpoint evaluation. Primary outcome measures will include success at gaining a competitive job, total hours of competitive employment, and neuropsychological measures of cognition.

DETAILED DESCRIPTION:
Background Information:

The Individual Placement and Support (IPS) program is an evidence-based vocational rehabilitation services that assist individuals with mental illness or significant mental health concerns gain and maintain competitive employment in the community. Unemployment rates among people with mental illness are high, even though most people with serious mental illness want to work.

Fraser Health provides IPS services to approximately 350 MHSU clients per year in six communities. The IPS strategy helps about 55% of clients find competitive jobs, but almost half (45%) fail to find work. Among those who fail to find employment, cognitive dysfunction is often a significant problem.

Cognitive remediation therapy (CRT) is an evidence-based, psychological treatment for the neurocognitive deficits seen in patients with severe mental illness. CRT targets cognitive functioning with the goal of improving role functioning in daily life. When compared with employment intervention alone, programs that incorporate CRT have shown a variety of vocational benefits, (e.g., more likely to work, held more jobs, worked more weeks, and earned more in wages) that are maintained even at a 3-year follow-up. CRT targeted to clients who have not been successful with IPS is efficient: non-responders improved employment outcome with a number needed-to-treat (NNT) of 4 over a two-year period.

Cognitive remediation (CRT) improves thinking skills and work functioning. CRT provides specific training modules and exercises that target thinking skills known to be impaired in severe mental illness. For example, working memory and cognitive flexibility are trained through real-world exercises that teach clients to organize and manage time, focus their attention, consider errors and their consequences, control answers and plan ahead. These skills are important to be successful in obtaining and maintaining employment.

Purpose of Study:

The primary purpose of this study is to assess, for people with serious mental illness who have failed to find employment despite three months of support in the IPS program, the effects of 12 weeks of cognitive remediation therapy (CRT) on subsequent employment outcomes while they continue to receive IPS employment-support services. Hypothesis:

The first hypothesis is that adding CRT for those who have not found employment by 3 months in the program will result in better competitive work outcomes, compared to those who continue IPS alone. The second hypothesis is that participants receiving CRT will improve more in cognitive functioning than those who did not receive CRT training. The third hypothesis is that symptom severity will be related to work outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 19-60 years old
* Enrolled in the IPS program for at least 3 months
* Clinically stable (no changes to psychiatric medication and psychiatric hospitalization in the 30 days prior to intake)

Exclusion Criteria:

* History of traumatic brain injury
* Neurological disorder
* Developmental disability
* Difficulty understanding written and spoken English

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Employment Outcomes | 90 days
  The number of hours client worked in the past 90 days.

SECONDARY OUTCOMES:
Cognitive Functioning | 90 minutes
  Cognitive functioning will be measured using the Matrics Consensus Cognitive Battery. The MCCB has 10 tests that measures 7 cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. Raw scores will be converted to T-score for each domain. T-score has a mean of 50 and a standard deviation of 10.
Psychiatric Symptoms | 2 weeks
  Brief Psychiatric Rating Scale. The BPRS is a semi-structured interview of psychiatric symptoms over the past 2 weeks. There are 24 items rated from 1 to 7 with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: David Erickson, PhD, Principal Investigator — Fraser Health
Locations (1):
- Fraser Health: Royal Columbian Hospital, New Westminster, British Columbia, Canada

REFERENCES:
- [Background] Marshall T, Goldberg RW, Braude L, Dougherty RH, Daniels AS, Ghose SS, George P, Delphin-Rittmon ME. Supported employment: assessing the evidence. Psychiatr Serv. 2014 Jan 1;65(1):16-23. doi: 10.1176/appi.ps.201300262. PMID 24247197
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] McGurk SR, Mueser KT. Cognitive functioning, symptoms, and work in supported employment: a review and heuristic model. Schizophr Res. 2004 Oct 1;70(2-3):147-73. doi: 10.1016/j.schres.2004.01.009. PMID 15329293
- [Background] McGurk SR, Mueser KT, Feldman K, Wolfe R, Pascaris A. Cognitive training for supported employment: 2-3 year outcomes of a randomized controlled trial. Am J Psychiatry. 2007 Mar;164(3):437-41. doi: 10.1176/ajp.2007.164.3.437. PMID 17329468
- [Background] McGurk SR, Mueser KT, Xie H, Welsh J, Kaiser S, Drake RE, Becker DR, Bailey E, Fraser G, Wolfe R, McHugo GJ. Cognitive Enhancement Treatment for People With Mental Illness Who Do Not Respond to Supported Employment: A Randomized Controlled Trial. Am J Psychiatry. 2015 Sep 1;172(9):852-61. doi: 10.1176/appi.ajp.2015.14030374. Epub 2015 May 22. PMID 25998278
- [Background] Bell MD, Zito W, Greig T, Wexler BE. Neurocognitive enhancement therapy with vocational services: work outcomes at two-year follow-up. Schizophr Res. 2008 Oct;105(1-3):18-29. doi: 10.1016/j.schres.2008.06.026. Epub 2008 Aug 19. PMID 18715755
- [Background] Kurtz MM, Wexler BE, Fujimoto M, Shagan DS, Seltzer JC. Symptoms versus neurocognition as predictors of change in life skills in schizophrenia after outpatient rehabilitation. Schizophr Res. 2008 Jul;102(1-3):303-11. doi: 10.1016/j.schres.2008.03.023. Epub 2008 May 20. PMID 18495433